CLINICAL TRIAL: NCT06633172
Title: Laparoscopic Ventral Mesh Rectopexy Versus Trans-vaginal Repair in Management of Anterior Rectocele; a Randomized Controlled Trial.
Brief Title: Laparoscopic Ventral Mesh Rectopexy Versus Trans-vaginal Repair for Anterior Rectocele.
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmad Sakr, principal investigator, Mansoura University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11111
Record Dates: First submitted 2024-10-04; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Rectocele; Anterior Rectocele
Keywords: transvaginal repair; ventral mesh rectopexy; laparoscopic
MeSH Terms: conditions — Rectocele

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- laparoscopic ventral mesh rectopexy (Active Comparator): performing laparoscopic ventral mesh rectopexy for group of patients to find out its efficacy
  Interventions: Procedure: laparoscopic ventral mesh rectopexy
- Trans vaginal repair (Active Comparator): performing trans vaginal repair for the 2nd group to find out its efficacy.
  Interventions: Procedure: Trans vaginal repair

INTERVENTIONS:
Procedure: laparoscopic ventral mesh rectopexy — performing ventral mesh rectopexy via laparoscopic surgery to correct the anterior rectocele.
  Other Names: VMR; ventral mesh rectopexy
  Arms: laparoscopic ventral mesh rectopexy
Procedure: Trans vaginal repair — performing repair of the rectocele through the recto vaginal septum repair.
  Other Names: TVR
  Arms: Trans vaginal repair

SUMMARY:
This study aims to compare the effect of laparoscopic ventral mesh rectopexy versus trans vaginal repair in management of anterior rectocele in females regarding functional outcomes.

DETAILED DESCRIPTION:
Rectocele is the protrusion of the anterior wall of the rectum into the vaginal lumen through the rectovaginal fascia and posterior vaginal wall. Symptomatic rectocele affects postmenopausal women and causes obstructed defecation Significant rectal emptying difficulties, straining at defecation, manually assisted defecation, the need for perineal or vaginal digitation, and local symptoms such as vaginal bulging and pelvic heaviness in 30-70% of cases have been described as symptoms of rectocele .

Constipation can be managed with dietary measures, laxatives, and biofeedback training , which can be beneficial for patients with modest symptoms. Surgical treatment is recommended if conservative treatment fails to alleviate symptoms . However, some patients may be left with constipation, fecal incontinence, incomplete bowel evacuation, or sexual dysfunction despite the correction of the anatomical defect. The selection of patients for surgical intervention for symptomatic rectocele remains a matter of debate.

There is still a controversy between abdominal approaches and the transanal, transperineal, and transvaginal approaches as the optimal surgical approach to treat complex rectocele. While the latter is preferred by gynecologists, the former has increased in popularity among colorectal surgeons, aided in part by the growing interest in minimally invasive surgery.

This study aimed to evaluate the outcome of LVMR in comparison with TVR of anterior rectocele regarding the improvement in constipation score and sexual-related quality of life, surgical outcomes and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 30 and 60 years, presented with symptomatic rectocele with failed conservative treatments.
* anterior rectocele larger than 3 cm in size with retention of the contrast in the rectocele on defecography.
* excessive straining, sense of incomplete evacuation, the need for digital manipulation during defecation, or dyspareunia.

Exclusion Criteria:

* significant urinary manifestations due to anterior vaginal wall prolapse.
* patients with recurrent rectocele
* complete external rectal prolapse
* isolated anismus
* connective tissue disease
* patients with slow-transit constipation
* fecal incontinence (FI), or abnormal thyroid function.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Improvement of constipation | 6 month to 1 year
  The primary outcome of the study was the absolute decline in constipation score(Cleveland clinic constipation score). This score is composed of 8 questions. Score ranges from 0 to 32. The lowest score is 0 which means no constipation, while the highest is 32 which means worsening of the constipation. So, the decline in the score means improving of the constipation.

SECONDARY OUTCOMES:
improvement of sexual function | 6 month to 1 year
  improvement in sexual function in the form of Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire(PISQ- 12). PISQ-12 score is composed of 3 domains with total score of 48. It ranges from 0 to 48. The higher the score, the better the sexual outcome.
  Other 2ry outcomes include: Operative time in minutes, time of wound healing in days and the postoperative complication in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Sakr, Phd, Principal Investigator — Mansoura University Hospital
Locations (1):
- Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sanad A, Sakr A, Elfeki H, Omar W, Thabet W, Fouda E, Abdallah E, Elbaz SA. Outcomes of laparoscopic ventral mesh rectopexy versus trans-vaginal repair in management of anterior rectocele, a randomized controlled trial. Tech Coloproctol. 2025 May 27;29(1):125. doi: 10.1007/s10151-025-03145-z. PMID 40423835